CLINICAL TRIAL: NCT00188825
Title: A Randomized, Double Blind, Placebo Controlled Study Comparing Simulect Plus Standard Immunosuppression to Standard Immunosuppression Alone for the Prevention of Acute Rejection and Bronchiolitis Obliterans Syndrome in Bilateral Lung and Single Lung Transplant Patients
Brief Title: Study Comparing Simulect Plus Standard Immunosuppression to Standard Immunosuppression Alone for the Prevention of Acute Rejection and Bronchiolitis Obliterans in Lung Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCHI621AES05
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: COPD; Emphysema; Alpha-1 Antitrypsan Deficiency
Keywords: Lung; Transplant; Rejection; BOS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Rejection, Psychology | interventions — Basiliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- basiliximab (Experimental)
  Interventions: Drug: basiliximab
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo
  Arms: placebo
Drug: basiliximab
  Arms: basiliximab

SUMMARY:
The study will evaluate the efficacy and safety of basiliximab Vs placebo as induction therapy combined with standard triple immunosuppression therapy, in the prevention of acute rejection episodes and prevention of Bronchiolitis Obliterans Syndrome.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of basiluximab for the prevention of acute allograft lung rejection when used in addition to Neoral, corticosteroids and azathioprine. Acute rejection episodes will be evaluated during the first 6 months post-transplant. Bronchiolitis obliterans syndrome (BOS) will be evaluated at the end of 1 year after transplant and at additional follow-up visits at 2 and 3 years after transplant.

ELIGIBILITY:
Inclusion criteria

* Male or female recipients of a first bilateral or single lung or lobar allograft who are suitable to receive Neoral/ corticosteroids/ azathioprine/ and Basiliximab (Simulect).
* Patients greater than 18 years of age.
* Patients capable of understanding the purposes and risks of the study and who have given informed written consent.

Exclusion Criteria:

* Patients who require immunosuppressive therapy other than the study medications.
* Patients participating in another (investigational) drug trial or who have participated in such a study within 30 days prior to transplantation.
* Pregnant mothers, nursing women.
* Women unwilling to use adequate contraception during and for 3 months after receiving study drug.
* Patients receiving or requiring other investigational drugs, except antibiotics.
* Patients with current or past peak panel reactive antibody levels of 25% or greater.
* Patients with malignancy or history of malignancy other than successfully treated non-metastatic basal cell or squamous cell carcinoma of the skin.
* Patients with any form of substance abuse or psychiatric disorder which, in the opinion of the investigator, might invalidate patient communication with the clinician(s).
* Patients who have previously received Simulect.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who experience one or more acute allograft rejections in the first six months of treatment.

SECONDARY OUTCOMES:
The proportion of patients who experience one or more acute allograft rejections by 1 year post-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Waddell, MD FRCSC, Principal Investigator — University Health Network, Toronto; Cecilia Chaparro, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada